CLINICAL TRIAL: NCT00819715
Title: Electrogastrography in Small for Gestational Age Preterm Infants Compared to Appropriate for Gestational Age Infants
Brief Title: Electrogastrography in Small for Gestational Age Preterm Infants
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Mrs. Leah Cohen, Meir Medical Center
Other Study IDs: 0244-07-MMC
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2009-06

CONDITIONS: Premature Birth
Keywords: Preterm infants; small for gestational age; electrogastrography
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Small for gestational age preterm infants
- 2: Appropriate for gestational preterm infants

SUMMARY:
The purpose of this study is to determine whether small for gestational preterm infants, have delayed or decrease gastric motility compared to appropriate for gestational age preterm infants.

ELIGIBILITY:
Inclusion Criteria:

1. preterm infants 32-37 weeks' gestation
2. No sepsis or ventilation
3. Feeding orally or with NG tube.
4. Age <48 h to be included

Exclusion Criteria:

1. GE reflux
2. Medication that affect gastric motility

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants >31 weeks, - 37 weeks , healthy, on enteralfeeds
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
EGG compatible with age | day 1 and day 7 after birth

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Arnon, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Neonatal Department,Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Result] Liang J, Co E, Zhang M, Pineda J, Chen JD. Development of gastric slow waves in preterm infants measured by electrogastrography. Am J Physiol. 1998 Mar;274(3):G503-8. doi: 10.1152/ajpgi.1998.274.3.G503. PMID 9530151